CLINICAL TRIAL: NCT00498433
Title: Part 1: An Open Label Pilot Study to Determine Interstitial and Tissue Concentrations of Aliskiren and Effects on the Renin- Angiotensin System (RAS) in Fat and Skeletal Muscle of Hypertensive Patients With Abdominal Obesity. Part 2: A Randomized, Double Blind, 12-weeks Parallel Group Study to Compare Effects of Aliskiren 300 mg and Amlodipine 5 mg on the RAS and Lipid/Carbohydrate Metabolism in Fat and Skeletal Muscle of Hypertensive Patients With Abdominal Obesity
Brief Title: Effects of Aliskiren and Amlodipine on the Renin-Angiotensin System (RAS) and Lipid/Carbohydrate Metabolism in Obese Patients With Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination resulted from interim analysis of the ALTITUDE trial
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2238
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Results first posted 2013-10-24 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension; Abdominal Obesity
Keywords: Aliskiren; Renin-Angiotensin System (RAS); Hypertension; Abdominal obesity
MeSH Terms: conditions — Hypertension; Obesity, Abdominal | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Experimental): Part 1: After a 1-2 weeks initial washout period, all eligible patients underwent a two week placebo run-in phase (period 1) consisting of treatment with one tablet of placebo to aliskiren once daily (o.d.). This was followed by a 4 week treatment phase (period 2) consisting of treatment with 300 mg aliskiren o.d..
  Part 2: Eligible randomized patients in this arm received aliskiren 300 mg tablet o.d. and amlodipine placebo capsule o.d. for 12 weeks.
  Interventions: Drug: Aliskiren; Drug: Placebo of Aliskiren; Drug: Placebo of amlodipine
- Amlodipine (Active Comparator): Part 1: After aliskiren treatment (period 2), each patient was entered into a second washout period (4 weeks) during which blood pressure was required to be ≤ 140/90 mmHg. If blood pressure exceeded 140/90 mmHg on two consecutive days (home monitoring) and was confirmed at the study center, the patient was entered into the amlodipine treatment period (period 3). In period 3, all patients received 5 mg amlodipine o.d.. The length of the amlodipine period varied from 4 to 7 weeks.
  Part 2: Eligible patients randomized to part 2 received amlodipine 5 mg o.d. and aliskiren placebo for 12 weeks
  Interventions: Drug: Amlodipine; Drug: Placebo of Aliskiren

INTERVENTIONS:
Drug: Aliskiren — 300 mg tablet once daily
  Other Names: SPP100
  Arms: Aliskiren
Drug: Amlodipine — 5 mg capsule once daily
  Arms: Amlodipine
Drug: Placebo of Aliskiren — Matching placebo of aliskiren 300 mg tablet
Drug: Placebo of amlodipine — Matching placebo of amlodipine 5 mg capsule
  Arms: Aliskiren

SUMMARY:
Part 1 determined: aliskiren, amlodipine and angiotensin II concentrations in interstitial fluid of fat and skeletal muscle; aliskiren and angiotensin II concentrations, and renin activity and concentration in fat and skeletal muscle tissues (biopsies); aliskiren, amlodipine and angiotensin II concentrations, and renin activity and concentration in plasma.

Part 2 investigated the potential for aliskiren to modulate renin-angiotensin-aldosterone system (RAAS) activity, and lipid/carbohydrate metabolism in adipose and skeletal muscle tissue in obese patients with hypertension in comparison to amlodipine.

ELIGIBILITY:
Inclusion criteria:

PART 1:

* Male and female patients 20 to 65 years of age with a diagnosis of hypertension and with abdominal obesity (waist circumference ≥ 102 cm in men and ≥ 88 cm in women)
* For patients with a history of treated hypertension, mean sitting systolic blood pressure (msSBP)/ mean sitting diastolic blood pressure (msDBP) had to be ≥ 120/80 mmHg and ≤ 160/100 mm Hg. For patients with newly diagnosed, untreated hypertension msSBP/msDBP had to be ≥ 135/85 mmHg and ≤ 160/100 mm Hg
* Pulse rate 40 - 90 bpm

PART 2:

* Male and female patients 18 to 65 years of age , with a diagnosis of hypertension and with abdominal obesity (waist circumference ≥ 102 cm in men and ≥ 88 cm in women)
* Systolic and diastolic blood pressure and pulse rate were assessed after the patient had rested for at least five (5) minutes. Vital signs had to be within the following ranges:

  1. Patients with history of treated hypertension: msSBP/msDBP ≥ 135/85 mmHg and < 160/100 mmHg at baseline
  2. Patients with newly diagnosed, untreated hypertension: msSBP/msDBP ≥ 135/85 mmHg and < 160/100 mmHg at screening and baseline.

Exclusion criteria:

PART 1

* Hypertension Grade 2 (msSBP ≥ 160 mmHg) or Grade 3 (msDBP ≥ 110 mmHg and/or msSBP ≥ 180 mmHg) WHO classification
* Current treatment with three or more antihypertensive drugs.

PART 2

* Hypertension Grade 2 (msSBP ≥ 160 and/or msDBP ≥ 100 mmHg).
* Current treatment with three or more antihypertensive drugs.

Other protocol-defined inclusion/exclusion criteria applied

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (2):
- Germany (2):
  - Novartis Investigative Site, Buch
  - Novartis Investigative Site, Hanover

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 46 patients entered into the study; 10 patients in part 1 received study drug. 36 patients enrolled into part 2 and and 16 patients received study drug.
Groups:
- Placebo: Part 1, Period 1: After a 1-2 weeks initial washout period, all eligible patients underwent a two week placebo run-in phase.
  Part 2, Period 1: After confirming study eligibility based on inclusion and exclusion criteria, patients underwent a two week single-blind placebo run-in phase.
- Aliskiren: Part 1 , Period 2: All eligible patients received 4 week treatment of 300 mg aliskiren o.d..
  Part 2, Double Blind Period: Eligible randomized patients received aliskiren 300 mg tablet o.d. and amlodipine placebo capsule o.d. for 12 weeks
- Amlodipine: Part 1, Period 3: All patients received 5 mg amlodipine o.d.. The length of the amlodipine period varied from 4 to 7 weeks.
  Part 2, Double Blind Period: Eligible randomized patients received amlodipine 5 mg o.d. and aliskiren placebo o.d. for 12 weeks
Period: Part 1, Period 1:Placebo Run-in(2 Weeks)
Arm/Group | Placebo | Aliskiren | Amlodipine
Started | 10 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part 1, Period 2: Aliskiren (4 Weeks)
Arm/Group | Placebo | Aliskiren | Amlodipine
Started | 0 | 10 | 0
Completed | 0 | 10 | 0
Not Completed | 0 | 0 | 0
Period: Part 1, Period 3: Amlodipine (4-8 Weeks)
Arm/Group | Placebo | Aliskiren | Amlodipine
Started | 0 | 0 | 10
Completed | 0 | 0 | 10
Not Completed | 0 | 0 | 0
Period: Part 2: Placebo Run-in (2 Weeks)
Arm/Group | Placebo | Aliskiren | Amlodipine
Started | 36 | 0 (For part 2, this arm belongs to randomized, double blind period.) | 0 (For part 2, this arm belongs to randomized, double blind period.)
Completed | 16 | 0 | 0
Not Completed | 20 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Abnormal laboratory value | 2 | 0 | 0
Not completed — Abnormal test procedure | 15 | 0 | 0
Not completed — Administrative problems | 1 | 0 | 0
Period: Part 2: Double Blind (12 Weeks)
Arm/Group | Placebo | Aliskiren | Amlodipine
Started | 0 | 8 | 8
Completed | 0 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 1 : Baseline measures are on all patients.
  Part 2: Randomized population of double-blind period used for Baseline/Demographic measurements.
Groups:
- Part 1: Placebo/Aliskiren/Amlodipine: Part 1, Period 1: After a 1-2 weeks initial washout period, all eligible patients underwent a two week placebo run-in phase.
  Part 1 , Period 2: All eligible patients received 4 week treatment of 300 mg aliskiren o.d..
  Part 1, Period 3: All patients received 5 mg amlodipine o.d.. The length of the amlodipine period varied from 4 to 7 weeks.
- Part 2, Double Blind Period: Aliskiren: Eligible randomized patients received aliskiren 300 mg tablet o.d. and amlodipine placebo capsule o.d. for 12 weeks
- Part 2, Double Blind: Amlodipine: Eligible randomized patients received amlodipine 5 mg o.d. and aliskiren placebo o.d. for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine | Part 2, Double Blind Period: Aliskiren | Part 2, Double Blind: Amlodipine | Total
Number analyzed (Participants) | 10 | 8 | 8 | 26
Age, Continuous [Mean (Standard Deviation); unit: years]
  Part 1, Open Label | 46 (7.5) | NA (NA) — This arm is used for part 2, double blind period | NA (NA) — This arm is used for part 2, double blind period | 46 (7.5)
  Part 2, Double blind | NA (NA) — This arm is used for part 1, open label . | 46.0 (10.92) | 49.4 (10.53) | 47.7 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 8 | 6 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Aliskiren Concentrations From Interstitial Fluid (Microdialysis)at the End of Aliskiren Treatment Period
Description: Interstitial fluid was obtained from subcutaneous adipose and skeletal muscle tissues by microdialysis using the zero-flow method. Interstitial fluid was collected for measurements of drug concentrations on the last day of the aliskiren treatment periods (Day 42).
Time Frame: Day 42
Population: All patients who received at least one dose of study drug and had at least one post-baseline assessment of pharmacokinetics (PK)/ pharmacodynamics (PD) data were included in the data analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
ng/mL
  Adipose tissue | 2.38 (2.11)
  Skeletal muscle | 7.05 (4.24)

2. Primary Outcome: Part 1: Amlodipine Concentrations From Interstitial Fluid (Microdialysis) at the End of Amlodipine Treatment Period
Description: Interstitial fluid was obtained from subcutaneous adipose and skeletal muscle tissues by microdialysis using the zero-flow method. Interstitial fluid was collected for measurements of drug concentration on the last day of the amlodipine treatment periods (Day 98).
Time Frame: Day 98
Population: Zero flow concentrations from microdialysates could not be derived by linear regression because of missing data due to inadequate sample volumes.
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 0

3. Secondary Outcome: Part 2: Microdialysis Metabolic Analytes in Response to Insulin Modified Frequently Sampled Intravenous Glucose Test [IM-FSIGT]for Each Tissue (Adipose or Skeletal Muscle)
Time Frame: Day 14 and Day 98
Population: Total 40 completed subjects needed to have a power of 80% in detecting a significant difference between treatment groups. Due to early termination, the study was limited by a small sample size; hence, the planned analysis was not done.
Groups:
- Aliskiren: Part 2, Double Blind Period: Eligible randomized patients received aliskiren 300 mg tablet o.d. and amlodipine placebo capsule o.d. for 12 weeks
- Amlodipine: Part 2, Double Blind Period: Eligible randomized patients received amlodipine 5 mg o.d. and aliskiren placebo o.d. for 12 weeks
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Part 2: Change From Baseline in Official Blood Pressure
Time Frame: Placebo Baseline (Day 14), Active Treatment (Day 98)
Population: as for outcome 3
Groups:
- Aliskiren: Part 2, Double Blind: Eligible randomized patients received aliskiren 300 mg tablet o.d. and amlodipine placebo capsule o.d. for 12 weeks
- Amlodipine: Part 2, Double Blind: Eligible randomized patients received amlodipine 5 mg o.d. and aliskiren placebo o.d. for 12 weeks
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Part 2: Renin Activity and Concentration of Aliskiren and Amlodipine in Fat and Skeletal Muscle Interstitial Fluid
Time Frame: Placebo Baseline (Day 14), Active Treatment (Day 98)
Population: as for outcome 3
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Part 1: Angiotensin II Levels in Interstitial Fluid of Fat and Skeletal Muscle (Microdialysis) During Aliskiren Treatment Period
Description: Interstitial fluid was obtained from subcutaneous adipose and skeletal muscle tissues by microdialysis using the zero-flow method to determine Ang II concentration.
Time Frame: Day 42
Population: Due to technical limitations, zero flow concentrations could not be derived for Ang II.
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 0

7. Primary Outcome: Part 1: Angiotensin II Levels in Interstitial Fluid of Fat and Skeletal Muscle (Microdialysis) During Amlodipine Treatment Period
Description: as for outcome 6
Time Frame: Day 98
Population: Due to technical limitations, zero flow concentrations could not be derived for Ang II.
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 0

8. Primary Outcome: Part 1: Aliskiren Concentrations From Tissue at the End of Aliskiren Treatment Period
Description: Biopsies were taken from abdominal adipose and skeletal muscle tissue to determine aliskiren concentration. Tissue biopsy samples for drug concentrations analyses were taken on the last day of the aliskiren treatment periods (Day 42).
Time Frame: Day 42
Population: All patients who received at least one dose of study drug and had at least one post-baseline assessment of pharmacokinetics data were included in the data analysis.
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 9
ng/g
  Adipose tissue (n=6) | 29.05 (16.71)
  Skeletal muscle (n=9) | 107.32 (68.64)

9. Primary Outcome: Part 1: Angiotensin II Levels From Tissue During Aliskiren Treatment Period
Description: Biopsies were taken from abdominal adipose and skeletal muscle tissue to determine Ang II concentration.
Time Frame: Day 42
Population: More than 50% of the biopsy samples over all time points were either below lower limit of quantification (LLOQ) or not received.
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 0

10. Primary Outcome: Part 1: Renin Activity and Concentrations From Adipose and Skeletal Tissues During Aliskiren Treatment Period
Time Frame: Day 42
Population: Renin activity and concentration from adipose tissue and skeletal muscles were all below lower limitation of quantification (LLOQ) at all time points.
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 0

11. Primary Outcome: Part 1: Aliskiren Concentrations From Plasma at the End of Aliskiren Treatment Period
Description: Plasma samples were obtained for measurement of aliskiren or amlodipine concentrations. All blood samples were taken by an indwelling cannula inserted in a forearm vein or direct venipuncture. The plasma samples for drug concentrations analyses were taken on the last day of the aliskiren treatment periods (Day 42).
Time Frame: Day 42
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
ng/mL | 8.38 (4.41)

12. Primary Outcome: Part 1: Amlodipine Concentrations From Plasma at the End of Amlodipine Treatment Period
Description: Plasma samples were obtained for measurement of aliskiren or amlodipine concentrations. All blood samples were taken by an indwelling cannula inserted in a forearm vein or direct venipuncture. The plasma samples for drug concentrations analyses were taken on the last day of the amlodipine treatment periods (Day 98).
Time Frame: Day 98
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
ng/mL | 7.78 (3.61)

13. Primary Outcome: Part 1: Angiotensin II Levels in Plasma During Aliskiren Treatment Period
Description: as for outcome 6
Time Frame: Day 42
Population: All patients who received at least one dose of study drug and had at least one post-baseline assessment of pharmacodynamic data were included in the data analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: fmol/mL
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
fmol/mL | 0.534 [0.223 to 1.28]

14. Primary Outcome: Part 1: Angiotensin II Levels in Plasma During Amlodipine Treatment Period
Description: as for outcome 6
Time Frame: Day 98
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: fmol/mL
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
fmol/mL | 2.20 [0.88 to 5.51]

15. Primary Outcome: Part 1: Renin Concentrations From Plasma During Aliskiren Treatment Period
Description: Renin concentrations from plasma were measured as: plasma renin concentration (PRC), prorenin concentration and total renin concentration (renin + prorenin concentration).
Time Frame: Day 42
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
pg/mL
  Plasma Renin Concentration | 22.29 [8.98 to 55.32]
  Total Renin Concentration | 89.9 [52.4 to 154.2]
  Prorenin Concentration | 62.1 [40.2 to 96.0]

16. Primary Outcome: Part 1: Renin Concentrations From Plasma During Amlodipine Treatment Period
Description: Renin concentrations from plasma were measured as plasma renin concentration (PRC), prorenin concentration and total renin concentration (renin + prorenin concentration).
Time Frame: Day 98
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
pg/mL
  Plasma Renin Concentration | 7.36 [4.24 to 12.80]
  Total Renin Concentration | 66.3 [49.8 to 88.2]
  Prorenin Concentration | 57.9 [44.1 to 76.1]

17. Primary Outcome: Part 1: Renin Activity From Plasma During Aliskiren Treatment Period
Description: Plasma Renin activity (PRC) was measured by a trapping PRA (tPRA) assay.
Time Frame: Day 42
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: ng/nl/h
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
ng/nl/h | 0.145 [0.055 to 0.386]

18. Primary Outcome: Part 1: Renin Activity From Plasma During Amlodipine Treatment Period
Description: Plasma renin activity (PRC) was measured by a trapping PRA (tPRA) assay.
Time Frame: Day 98
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: ng/nl/h
Arm/Group | Part 1: Placebo/Aliskiren/Amlodipine
Number analyzed (Participants) | 10
ng/nl/h | 0.670 [0.269 to 1.672]

19. Primary Outcome: Part 2: Change From Baseline in Angiotensin II Levels in Interstitial Fluid of Fat and Skeletal Muscle (Microdialysis) During Double Blind Treatment Period
Description: as for outcome 6
Time Frame: Placebo Baseline (Day 14), Active Treatment (Day 98)
Population: as for outcome 3
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Part 2: Change From Baseline in Plasma Angiotensin II Levels During Double Blind Treatment Period
Description: Plasma Ang II was measured prior to and 1 hour after the Insulin modified-frequently sampled intravenous glucose tolerance test (IM-FSIGT) during placebo treatment (Days 14) and active treatment(Day 98).
Time Frame: Placebo Baseline (Day 14), Active Treatment (Day 98)
Population: as for outcome 3
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Part 2: Plasma Renin Activity (PRA) Concentration During Double Blind Treatment Period
Time Frame: Day 98
Population: as for outcome 3
Groups:
- Aliskiren: Part 2, Double Blind Period: Eligible randomized patients of this arm received aliskiren 300 mg tablet o.d. and amlodipine placebo capsule o.d. for 12 weeks
- Amlodipine: Part 2, Double Blind Period: Eligible randomized patients of this arm received amlodipine 5 mg o.d. and aliskiren placebo o.d. for 12 weeks
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Part 2: Plasma Renin Concentration (PRC) Levels During Double Blind Treatment Period
Time Frame: Day 98
Population: as for outcome 3
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Part 2: Change From Baseline in Peripheral Insulin Sensitivity in Response to Insulin Modified Frequently Sampled Intravenous Glucose Test [IM-FSIGT]for Each Tissue (Adipose or Skeletal Muscle)
Time Frame: Placebo Baseline (Day 14), Active Treatment (Day 98)
Population: as for outcome 3
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Part 2: Change From Baseline in Mitochondrial Mass in Subcutaneous Fat and Skeletal Muscle (Tissue Biopsies)
Time Frame: Placebo Baseline (Day 14), Active Treatment (Day 98)
Population: as for outcome 3
Arm/Group | Aliskiren | Amlodipine
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Part 2: Number of Participants With Reported Any Adverse Events, Serious Adverse Events and Death
Time Frame: 98 days
Population: The safety population consisted of all patients who received at least one dose of study drug with at least one post-baseline safety assessment. Patients were analyzed according to treatment received.
Measure: Number; unit: Participants
Groups:
- Placebo run-in: Part 2, Period 1, Placebo run-in phase: After confirming study eligibility based on inclusion and exclusion criteria, patients will undergo a two week single-blind placebo run-in phase.
- Amlodipine: Part 2, Double Blind: Eligible randomized patients of this arm received amlodipine 5 mg o.d. and aliskiren placebo o.d. for 12 weeks
Arm/Group | Placebo run-in | Aliskiren | Amlodipine
Number analyzed (Participants) | 36 | 8 | 8
Participants
  Adverse event | 9 | 2 | 3
  Serious Adverse Event | 1 | 0 | 0
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Description: The Safety Population consisted of all patients that received at least one dose of study drug with at least one post-baseline safety assessment.
  In Part 1 of the study, no events were reported in period 1 when patients received placebo.
Groups:
- Part 1: Aliskiren: All eligible patients received 4 week treatment of 300 mg aliskiren o.d..
- Part 1: Amlodipine: All patients received 5 mg amlodipine o.d.. The length of the amlodipine period varied from 4 to 7 weeks.
- Part 2: Placebo run-in Period: After confirming study eligibility based on inclusion and exclusion criteria, patients will undergo a two week single-blind placebo run-in phase.
- Part 2: Aliskiren: Eligible randomized patients of this arm received aliskiren 300 mg tablet o.d. and amlodipine placebo capsule o.d. for 12 weeks
- Part 2: Amlodipine: Double Blind Period: Eligible randomized patients of this arm received amlodipine 5 mg o.d. and aliskiren placebo o.d. for 12 weeks
Arm/Group | Part 1: Aliskiren | Part 1: Amlodipine | Part 2: Placebo run-in Period | Part 2: Aliskiren | Part 2: Amlodipine
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 1/36 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/10 | 3/10 | 1/36 | 2/8 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Aliskiren (N=10) | Part 1: Amlodipine (N=10) | Part 2: Placebo run-in Period (N=36) | Part 2: Aliskiren (N=8) | Part 2: Amlodipine (N=8)
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Aliskiren (N=10) | Part 1: Amlodipine (N=10) | Part 2: Placebo run-in Period (N=36) | Part 2: Aliskiren (N=8) | Part 2: Amlodipine (N=8)
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
IRRITABILITY (General disorders) | 0 | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 2 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
WEIGHT INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.